CLINICAL TRIAL: NCT00839930
Title: A Relative Bioavailability Study of 50 mg Cilostazol Tablets Under Fasting Conditions
Brief Title: Cilostazol 50 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: R04-099
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cilostazol (test) (Experimental): Cilostazol 50 mg Tablet (test) dosed in first period followed by Pletal® 50 mg Tablet (reference) dosed in second period
  Interventions: Drug: Cilostazol 50 mg Tablets
- Pletal® (reference) (Active Comparator): Pletal® 50 mg Tablet (reference) dosed in first period followed by Cilostazol 50 mg Tablet (test) dosed in second period.
  Interventions: Drug: Pletal®

INTERVENTIONS:
Drug: Cilostazol 50 mg Tablets — 1 x 50 mg, single-dose fasting
  Arms: Cilostazol (test)
Drug: Pletal® — 1 x 50 mg, single-dose tablet
  Arms: Pletal® (reference)

SUMMARY:
This study will compare the relative bioavailability (rate and extent of absorption) of 50 mg Cilostazol Tablets manufactured by TEVA Pharmaceuticals Industries Ltd. and distributed by TEVA Pharmaceuticals USA with that of PLETAL Tablets manufactured by Otsuka Pharmaceuticals Co., Ltd. for Otsuka America Pharmaceutical, Inc. following a single oral dose (1 x 50 mg tablet) in healthy adult subjects administered under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All volunteers selected for this study will be healthy men or women 18 years of age or older at the time of dosing. The volunteer's body mass index (BMI) is less than or equal to 30.
* Screening Procedures: Each volunteer will complete the screening process within 28 days prior to Period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.

Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory, and central nervous systems.

* The screening clinical laboratory procedures will include:

  * Hematology: hematocrit, hemoglobin, RBC count, WBC count with differential, platelet count;
  * Clinical Chemistry: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase.
  * HIV antibody and hepatitis B surface antigen and hepatitis C antibody screens;
  * Urinalysis: by dipstick; full microscopic examination if dipstick positive; and
  * Urine Drug Screen: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates, and phencyclidine;
  * Serum Pregnancy Screen (female volunteers only).
  * Follicle Stimulating Hormone (FSH; female subjects only): verify postmenopausal status
* If female and:

  * is postmenopausal for at least 1 year with postmenopausal status defined as: > 60 years of age and amenorrheic for at least one year; if 60 years of age or younger, must also have a serum FSH level >30 IU/L; or
  * is surgically sterile for at least 6 months (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

* Volunteers with a recent history of drug or alcohol addiction or abuse.
* Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators).
* Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Volunteers demonstrating a positive hepatitis B surface antigen screen or a reactive HIV antibody screen.
* Volunteers demonstrating a positive drug abuse screen when screened for this study.
* Female volunteers demonstrating a positive pregnancy screen.
* Female volunteers who are currently breastfeeding.
* Volunteers with a history of allergic response(s) to cilostazol or related drugs.
* Volunteers with a history of clinically significant allergies including drug allergies.
* Volunteers with a clinically significant illness during 4 weeks prior to Period I dosing (as determined by the clinical investigators).
* Volunteers who are currently using or report using tobacco products within 90 days prior to Period I dosing.
* Volunteers who have taken any drug known to induce or inhibit hepatic drug metabolism in the 30 days prior to Period I dosing.
* Volunteers who report donating greater than 150 mL of blood within 30 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
* Volunteers who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
* Volunteers who report receiving any investigational drug within 30 days prior to Period I dosing.
* Volunteers who report taking any prescription medication or nonprescription medication in the 14 days or 7 days, respectively, prior to Period I dosing with the exception of topical products without systemic absorption.
* Volunteers who have been on an abnormal diet during the 28 days prior to Period I dosing.
* Volunteers who report an intolerance or direct venipuncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-02; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Carlson, Pharm.D., Principal Investigator — PRACS Institute, Ltd.
Locations (2):
- United States (2):
  - PRACS Institute Ltd., East Grand Forks, Minnesota
  - PRACS Institute, Ltd., Fargo, North Dakota

RESULTS

PARTICIPANT FLOW:
Groups:
- Cilostazol (Test) First: Cilostazol 50 mg Tablets (test)dosed in first period followed by Pletal® 50 mg Tablets (reference) dosed in second period
- Pletal® (Reference) First: Pletal® 50 mg Tablets (reference) dosed in first period followed by Cilostazol 50 mg Tablets (test) dosed in second period
Period: First Intervention
Arm/Group | Cilostazol (Test) First | Pletal® (Reference) First
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Washout: 7 Days
Arm/Group | Cilostazol (Test) First | Pletal® (Reference) First
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Cilostazol (Test) First | Pletal® (Reference) First
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cilostazol (Test) First | Pletal® (Reference) First | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 6
  Male | 15 | 9 | 24
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 15 | 14 | 29
  Asian | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cilostazol: Cilostazol 50 mg Tablets (test)dosed in either period
- Pletal®: Pletal® 50 mg Tablets (reference) dosed in either period
Arm/Group | Cilostazol | Pletal®
Number analyzed (Participants) | 30 | 30
ng/mL | 376.46 (115.88) | 398.06 (108.07)
Statistical Analysis 1: Comparison: Cilostazol vs Pletal®; Test type: Non-Inferiority or Equivalence — Analysis of Variance (ANOVA) will be performed on the log-transformed AUC0-t, AUC0-inf and Cmax parameters; Geometric Test/Ref Ratio x 100 = 93.39, 90% CI [87.33 to 99.86] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cilostazol | Pletal®
Number analyzed (Participants) | 30 | 30
ng*h/mL | 5010.17 (1508.03) | 5176.83 (1435.42)
Statistical Analysis 1: Comparison: Cilostazol vs Pletal®; Test type: Non-Inferiority or Equivalence — Analysis of Variance (ANOVA) will be performed on the log-transformed AUC0-t, AUC0-inf and Cmax parameters; Geometric Test/Ref Ratio x 100 = 96.14, 90% CI [91.04 to 101.52] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cilostazol | Pletal®
Number analyzed (Participants) | 30 | 30
ng*h/mL | 4618.70 (1416.60) | 4745.22 (1370.01)
Statistical Analysis 1: Comparison: Cilostazol vs Pletal®; Test type: Non-Inferiority or Equivalence — Analysis of Variance (ANOVA) will be performed on log-transformed AUC0-t, AUC0-inf and Cmax parameters; Geometric Test/Ref Ratio x 100 = 96.64, 90% CI [92.13 to 101.37] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.